CLINICAL TRIAL: NCT05755503
Title: Toxicokinetics of Protein-bound Uremic Toxins in ESRD Patients
Status: Recruiting | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Ding Feng, professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: JYLJ202218
Record Dates: First submitted 2023-03-02; First posted 2023-03-06 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Uremic; Toxemia; Pharmacokinetics; Renal Dialysis
Keywords: Renal Dialysis; Uremic; Toxemia; Pharmacokinetics
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples;urine samples;dialysate samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IS modeling and validation group: Uremia patients receiving hemodialysis.This group was used to establish the IS three-compartment model and verify the accuracy and predictive value of the model

SUMMARY:
Protein-bound uremic toxins (PBUTs) are important uremic toxins, represented by indoxyl sulfate (IS), derived from the fermentation of dietary proteins by gut bacteria. The purpose of this study was to study the changes of IS in maintenance hemodialysis patients, and to construct a metabolic kinetics model of IS clearance. The model was then used to estimate the clearance rate of indoxyl sulfate by hemoperage, and to verify the application value of the model. This study intends to collect a series of serum, dialysate and urine samples from maintenance hemodialysis patients receiving high-throughput dialysis or hemodialysis filtration, so as to clarify the variation rule of IS during various blood purification treatments. Furthermore, a three-compartment model of dialysis IS metabolism kinetics was constructed according to the IS clearance of dialysis and residual kidney, and the above model was verified internally and externally. Finally, the model's fit and predictive value were validated in a group of MHD patients treated with HP without residual kidney.

DETAILED DESCRIPTION:
The results of this study are helpful to clarify the rules of clearance and metabolism of PBUTs in hemodialysis patients, and lay a foundation for exploring effective means of blood purification and drugs to eliminate PBUTs, so as to reduce the incidence and mortality of complications in uremia patients.

Hemodialysis parameter setting: Blood flow 250ml/min, high throughput dialysis mode, dialysis process lasted for 4h

Samples collection time point:Blood samples: before hemodialysis, 1h, 2h, 4h after hemodialysis, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h, 48h after hemodialysis.Dialysate samples: 1h, 1.5h, 2h, 3h, 4h after hemodialysis.Urine samples: 4h urine samples during hemodialysis.Hemoperfusion samples: before hemodialysis, 5min, 15min, 30min, 45min, 60min, 90min, 120min after hemodialysis.

The proposed model of IS toxicokinetics is a three-compartment model, in which the circulatory system is the central compartment, intertissue fluid is the fast equilibrium chamber, and cerebrospinal fluid, intracellular fluid, lymphatic fluid, etc. are the slow equilibrium chamber

ELIGIBILITY:
Inclusion Criteria:

1. Patients with maintenance hemodialysis were less than 85 years old and more than 18 years old, both male and female;
2. Regular hemodialysis for more than 3 months, using arteriovenous fistula hemodialysis;
3. Receiving high-throughput dialysis, HDF, and HP according to the conventional treatment regimen;
4. Adequate dialysis (Kt/V>1.2 within one month);
5. Keep your diet steady. Generally in good condition, have self-awareness, have a good understanding of their own illness and physical condition, and can communicate well with others;
6. Understand and sign the informed consent

Exclusion Criteria:

1. Patients with systemic or local severe infection;
2. Patients with severe anemia: Hb<60g/L;
3. Patients with hypoproteinemia: Alb<30g/L;
4. Patients with insufficient daily protein intake: nPCR>1.0g/kg/d;
5. Patients with malignant tumors;
6. Patients with severe cardiovascular and cerebrovascular diseases, such as unstable angina pectoris, malignant hypertension, persistent atrial fibrillation, abnormal Q-wave of electrocardiogram, or patients with acute myocardial infarction, stroke, or coronary stent implantation within 3 months;
7. Patients with severe hematopoietic system diseases, such as aplastic anemia, globin aplastic anemia, thrombocytopenic purpura, etc.;
8. Patients with severe digestive diseases, such as dysphagia, liver insufficiency, active gastrointestinal bleeding, intestinal obstruction, intestinal perforation, or previous subtotal gastrectomy, and other diseases that may affect digestion and absorption;
9. Pregnant women;
10. Participating in other clinical trials within one month or currently;
11. Researchers consider it inappropriate.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Uremia patients with maintenance hemodialysis in Shanghai ninth people's hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The blood concentration of IS | From the beginning of dialysis to 48 hours after dialysis
  The concentration of the free and protein-bound IS
The dialysate concentration of IS | Four hours of dialysis
  The concentration of the free and protein-bound IS
The urine concentration of IS | Four hours of dialysis
  The concentration of the free and protein-bound IS

SECONDARY OUTCOMES:
Dialytic clearance | Four hours of dialysis
  The total IS amount removed by dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Ding Feng, PhD, Study Director — Division of Nephrology,Shanghai Ninth People's Hospital
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maheshwari V, Thijssen S, Tao X, Fuertinger D, Kappel F, Kotanko P. A novel mathematical model of protein-bound uremic toxin kinetics during hemodialysis. Sci Rep. 2017 Sep 4;7(1):10371. doi: 10.1038/s41598-017-10981-z. PMID 28871178
- [Background] Meyer TW, Peattie JW, Miller JD, Dinh DC, Recht NS, Walther JL, Hostetter TH. Increasing the clearance of protein-bound solutes by addition of a sorbent to the dialysate. J Am Soc Nephrol. 2007 Mar;18(3):868-74. doi: 10.1681/ASN.2006080863. Epub 2007 Jan 24. PMID 17251385
- [Background] Esquivias-Motta E, Martin-Malo A, Buendia P, Alvarez-Lara MA, Soriano S, Crespo R, Carracedo J, Ramirez R, Aljama P. Hemodiafiltration With Endogenous Reinfusion Improved Microinflammation and Endothelial Damage Compared With Online-Hemodiafiltration: A Hypothesis Generating Study. Artif Organs. 2017 Jan;41(1):88-98. doi: 10.1111/aor.12704. Epub 2016 May 16. PMID 27182679
- [Background] Devine E, Krieter DH, Ruth M, Jankovski J, Lemke HD. Binding affinity and capacity for the uremic toxin indoxyl sulfate. Toxins (Basel). 2014 Jan 24;6(2):416-29. doi: 10.3390/toxins6020416. PMID 24469432